CLINICAL TRIAL: NCT03412734
Title: Is Chlorhexidine Vaginal Preparation Prior to Hysterectomy Superior to Iodine in Reducing Bacterial Count; a Randomized Controlled Trial
Brief Title: Vaginal Preparation Prior to Hysterectomy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The institutional review board recommended the study stop enrollment prior to achieving its initial sample size for patient safety.
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17-102
Record Dates: First submitted 2018-01-22; First posted 2018-01-26 (Actual); Results first posted 2020-11-18 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Hysterectomy
MeSH Terms: interventions — Chlorhexidine; Iodine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Chlorhexidine group (Experimental)
  Interventions: Drug: Chlorhexidine
- Iodine group (Active Comparator)
  Interventions: Drug: Iodine

INTERVENTIONS:
Drug: Chlorhexidine — Chlorhexidine preparation solutions
  Arms: Chlorhexidine group
Drug: Iodine — Iodine-based preparation solutions
  Arms: Iodine group

SUMMARY:
This is a randomized controlled trial to determine the influence of chlorhexidine gluconate surgical/topical antiseptic solutions on the bacterial environment of the vagina during hysterectomy and compare that to the effect of standard iodine-based preparations on the same.

DETAILED DESCRIPTION:
Postoperative infection remains the most common complication of surgical procedures in gynecology. Historically, 30-40% of patients undergoing a hysterectomy develop a post-operative infection. The initiation of antibiotic prophylaxis for appropriate surgical procedures was a significant advancement in the prevention of surgical site infection.

Antibiotic prophylaxis has been standardized and universally implemented. A remaining variable is the method of aseptic preparation of the vagina with substantial variation of technique being reported even within institutions.

The most recent Committee Opinion by the American College of Obstetricians and Gynecologists concludes there is insufficient evidence to render a strong recommendation for either povidone-iodine or chlorhexidine as the ideal agent for surgical preparation of the vagina and that further evidence is necessary.

Povidone-iodine solution has been considered the standard for aseptic surgical preparation of the vagina for decades and is the only solution approved by the FDA for vaginal use. There are however specific qualities of the solution that suggest it may be less than ideal for use in the vagina. More contemporary efforts have begun to focus on chlorhexidine as a more ideal agent for aseptic efforts in surgical preparation of the vagina.

The purpose of our study is to use a randomized controlled trial to determine if chlorhexidine gluconate surgical preparation maintains a lower rate of contamination to the surgical field.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing total vaginal, laparoscopic assisted vaginal, total laparoscopic, or robotic-assisted laparoscopic hysterectomy by a physician at Cincinnati Urogynecology Associates or Tri-State Gynecology Oncology TriHealth Inc.
* Concomitant procedures such as vaginal vault suspension, suburethral sling, cystoscopy, enterocele repair, anterior or posterior colporrhaphy, bilateral salpingectomy or salpingooophorectomy, staging procedures, lymph node sampling and other indicated procedures will be included
* English speaking
* Ability to provide consent

Exclusion Criteria:

* Unwillingness to participate in the study
* Non English speaking
* Patients that do not undergo a hysterectomy
* Reported allergy to iodine or chlorhexidine preparation solutions
* Patients undergoing planned debulking surgery for ovarian, fallopian tube or primary peritoneal cancers
* Current infection necessitating hysterectomy
* Active sepsis, pelvic abscess or pelvic inflammatory disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2018-05-18 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2020-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catrina Crisp, MD, Principal Investigator — TriHealth - Cincinnati Urogynecology Associates
Locations (1):
- Good Samaritan Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nugent RP, Krohn MA, Hillier SL. Reliability of diagnosing bacterial vaginosis is improved by a standardized method of gram stain interpretation. J Clin Microbiol. 1991 Feb;29(2):297-301. doi: 10.1128/jcm.29.2.297-301.1991. PMID 1706728
- [Derived] Hill AM, Pauls RN, Basil J, Tam T, Yook E, Shatkin-Margolis A, Kleeman S, Yeung J, Aldrich E, Crisp CC. Chlorhexidine Versus Iodine for Vaginal Preparation Before Hysterectomy: A Randomized Clinical Trial. Female Pelvic Med Reconstr Surg. 2022 Feb 1;28(2):77-84. doi: 10.1097/SPV.0000000000001066. PMID 34333502

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 6 patients were excluded (3 - not randomized at the day of surgery; 3 - missing study consent).
Groups:
- Chlorhexidine Group: Patients randomized to the Chlorhexidine group will undergo pre-surgical vaginal aseptic preparation using 4% Chlorhexidine preparation solutions.
- Iodine Group: Those patients randomized to the povidone-iodine group will have their pre-surgical vaginal aseptic preparation performed using 10% povidone-iodine solution.
Period: Overall Study
Arm/Group | Chlorhexidine Group | Iodine Group
Started | 47 | 41
Completed | 44 | 41
Not Completed | 3 | 0
Not completed — Incorrect labeling of samples | 2 | 0
Not completed — Exclusion criteria - patient receiving Flagyl for treatment | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chlorhexidine Group | Iodine Group | Total
Number analyzed (Participants) | 44 | 41 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (10.9) | 62.2 (11.6) | 59.8 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 41 | 85
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 42 | 39 | 81
  Black/African American | 2 | 1 | 3
  Asian | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 44 | 41 | 85
Bacterial Vaginosis (BV) positive [Count of Participants; unit: Participants] — Bacterial Vaginosis was identified through a modified Nugent method (Nugent RP et al. 1991), and Nugent score points was awarded based on three morphotypes:
  medium to large gram positive rods, small gram negative or variable rods, curved gram negative or variable rods.
  Each of these morphotypes was assigned a score based on their initial count, and the three morphotypes is then added, and any score >7 is consistent bacterial vaginosis, and a score <3 is normal flora.
  Participants | 12 | 18 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Contamination
Description: Contamination is defined as having >5000 bacteria within a culture
Time Frame: 90 minutes from initial preparation
Population: Use participants with cultures at 90 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Chlorhexidine Group | Iodine Group
Number analyzed (Participants) | 42 | 41
Participants | 20 | 35
Statistical Analysis 1: Comparison: Chlorhexidine Group vs Iodine Group; We hypothesized that chlorhexidine would have a lower bacterial count compared to iodine. Our sample size was calculated to be 71 patients per arm to detect a 22% difference in cultures defined as contaminated at 90 minutes from surgical preparation; Test type: Other; p < 0.001, Regression, Logistic — p-value is adjusted for baseline BV (Bacterial Vaginosis); Odds Ratio (OR) = 10.6, 95% CI 2-sided [3.02 to 37.34]

ADVERSE EVENTS:
Time Frame: 2 week post-op
Arm/Group | Chlorhexidine Group | Iodine Group
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/41
Other Adverse Events (participants affected / at risk) | 0/44 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-20): https://cdn.clinicaltrials.gov/large-docs/34/NCT03412734/Prot_SAP_000.pdf